CLINICAL TRIAL: NCT00216970
Title: Study of Arginine Metabolism and Nitric Oxide Formation in Relation to Glutamine Supply in Severely Burned Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ronald G. Tompkins, MD, ScD, Chief, Burn Service, Massachusetts General Hospital
Organization: National Institute of General Medical Sciences (NIGMS) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1999-P-008460; 5P50GM021700-28 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Burns
Keywords: parenteral nutrition; burn injury; stable isotopes; Arginine Metabolic Kinetics; Nitric Oxide Formation; Glutamine Metabolic Kinetics
MeSH Terms: conditions — Burns; Hyperphagia | interventions — Nutritional Support; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Patients will receive nutritional support in which the contents of arginine = 0, glutamate = 0 and proline = 0.
  Stable isotope tracer studies will be conducted to investigate the whole body protein metabolism and the utilization of arginine in critically ill burn patients.
  Interventions: Dietary Supplement: Alteration in nutritional support
- 2 (No Intervention): In arm 2 patients will receive nutritional support which will provide glutamine 0.5g/kg/day. Stable isotope tracer studies will be conducted to investigate the whole body protein metabolism and the utilization of arginine in critically ill burn patients.
  Interventions: Dietary Supplement: Alteration in nutritional support

INTERVENTIONS:
Dietary Supplement: Alteration in nutritional support — The subject is randomized into one of two groups - One receives TPN that does not have arginine, proline or glutamate. The other will receive TPN with extra glutamine. The subject takes part in 3 tracer studies while in the hospital. For each tracer study, the subject will receive a different randomly assigned diet. Blood and air are sampled and the patient receives a stable isotope after which the tests are repeated.
  Other Names: Dietary Supplement; Nutritional Evaluation

SUMMARY:
The purpose of the study is to understand the way the body uses amino acids and proteins in burned patient during the time they cannot eat normally. This study aims to understand the metabolism of the amino acid arginine in the body after burn injury. The results of this study will help determine the best composition of food needed during an acute burn injury so that body can more efficiently use the supplied nutrient for optimal burn wound healing and early recovery.

DETAILED DESCRIPTION:
The principle sources of plasma free arginine are (i) diet, (ii) release from protein breakdown and (iii) de novo synthesis directly from citrulline and the recycling of orthinine via the urea cycle. The major pathway of arginine disposal is i)oxidation via orthinine glutamate and subsequently the Tricarboxylic Acid (TCA) cycle and ii)via formation of nitric oxide. The latter pathway plays an important regulatory role in the body's response to stress and is significantly increased after burn injury.

Previous studies with burn patients show i)an increased rate of total arginine flux, ii)a limited rate of arginine de novo synthesis, and iii) an apparent increase in the rate of arginine catabolism as measured indirectly by increased orinthine oxidation. These changes render arginine a conditionally essential amino acid for burn patients. Studies have shown that feeding glutamine to healthy adults significantly alters the blood concentrations of urea cycle intermediates arginine, citrulline and orthinine. Therefore, we hypothesize that the availability of arginine can be improved in the burn patient by supplementing total parenteral nutrition (TPN) support with glutamine.

Using stable isotope tracer studies our specific aims are:

1. To explore the dynamic aspects of arginine and citrulline metabolism. There will be an emphasis on arginine disposal via oxidation and urea nitrogen formation via nitric oxide production.
2. To explore the effect of a) depleting arginine and its immediate precursors proline and glutamine, and b)glutamine supplementation on the metabolic pathways of burn patients.
3. To estimate the rate of nitric oxide (NO) formation in burn patients using arginine and citrulline tracers

ELIGIBILITY:
Inclusion Criteria:

* Burn patients being treated at MGH Burn Unit with one or more of the following criteria: 1) >=5% TBSA; 2) inhalation injury; or 3) resting energy expenditure (REE) of >15% of the predicted Basal Metabolic Rate using the Harris-Benedict equation.
* Must be receiving total parenteral nutrition in the course of their treatment.

Exclusion Criteria:

* Patients with thyroid disease
* Patients who are not hemodynamically stable or show unstable vital signs
* Patients at the stage of major organ failure, e.g. renal and/or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 1997-08; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
This is a nutritional study. The primary outcome is to measure the protein kinetics of amino acid metabolism. Fate will be determine from measurements of subject blood and air samples. | 18 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Tompkins, MD, ScD, Principal Investigator — MGH, Shriner's Burn Hospital -Boston
Locations (1):
- MGH Burn Unit, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tharakan JF, Yu YM, Zurakowski D, Roth RM, Young VR, Castillo L. Adaptation to a long term (4 weeks) arginine- and precursor (glutamate, proline and aspartate)-free diet. Clin Nutr. 2008 Aug;27(4):513-22. doi: 10.1016/j.clnu.2008.04.014. Epub 2008 Jun 30. PMID 18590940
- [Background] Yu YM, Ryan CM, Castillo L, Lu XM, Beaumier L, Tompkins RG, Young VR. Arginine and ornithine kinetics in severely burned patients: increased rate of arginine disposal. Am J Physiol Endocrinol Metab. 2001 Mar;280(3):E509-17. doi: 10.1152/ajpendo.2001.280.3.E509. PMID 11171607
- [Background] Yu YM, Ryan CM, Burke JF, Tompkins RG, Young VR. Relations among arginine, citrulline, ornithine, and leucine kinetics in adult burn patients. Am J Clin Nutr. 1995 Nov;62(5):960-8. doi: 10.1093/ajcn/62.5.960. PMID 7572742
- [Background] Castillo L, DeRojas-Walker T, Yu YM, Sanchez M, Chapman TE, Shannon D, Tannenbaum S, Burke JF, Young VR. Whole body arginine metabolism and nitric oxide synthesis in newborns with persistent pulmonary hypertension. Pediatr Res. 1995 Jul;38(1):17-24. doi: 10.1203/00006450-199507000-00004. PMID 7478791
- [Background] Yu YM, Young VR, Castillo L, Chapman TE, Tompkins RG, Ryan CM, Burke JF. Plasma arginine and leucine kinetics and urea production rates in burn patients. Metabolism. 1995 May;44(5):659-66. doi: 10.1016/0026-0495(95)90125-6. PMID 7752916